CLINICAL TRIAL: NCT05068284
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of ABBV-154 in Subjects With Moderately to Severely Active Crohn's Disease (CD): AIM-CD
Brief Title: A Study to Evaluate Adverse Events and Change in Disease Activity in Participants Between 18 to 75 Years of Age Treated With Intravenous (IV) Infusion and Subcutaneous (SC) Injections of ABBV-154 for Moderately to Severely Active Crohn's Disease
Acronym: AIM-CD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: M20-371; 2021-002869-18 (EudraCT Number)
Record Dates: First submitted 2021-09-27; First posted 2021-10-05 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; ABBV-154
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (10):
- Induction Phase: ABBV-154 Randomized Dose A (Experimental): Varying doses of ABBV-154 as described in the protocol.
  Interventions: Drug: ABBV-154
- Induction Phase: ABBV-154 Randomized Dose B (Experimental): Varying doses of ABBV-154 as described in the protocol.
  Interventions: Drug: ABBV-154
- Induction Phase: ABBV-154 Randomized Dose C (Experimental): Varying doses of ABBV-154 as described in the protocol.
  Interventions: Drug: ABBV-154
- Induction Phase: ABBV-154 Randomized Dose D (Experimental): Varying doses of ABBV-154 as described in the protocol.
  Interventions: Drug: ABBV-154; Drug: Placebo
- Induction Phase: Randomized Placebo (Placebo Comparator): Fixed dose placebo as described in the protocol.
  Interventions: Drug: Placebo
- Re-Induction Phase: ABBV-154 Randomized Dose A (Experimental): Varying doses of ABBV-154 as described in the protocol.
  Interventions: Drug: ABBV-154
- Re-Induction Phase: ABBV-154 Randomized Dose B (Experimental): Varying doses of ABBV-154 as described in the protocol.
  Interventions: Drug: ABBV-154
- Maintenance Phase: ABBV-154 Randomized Dose A (Experimental): Fixed dose ABBV-154 every other week.
  Interventions: Drug: ABBV-154
- Maintenance Phase: ABBV-154 Randomized Dose B (Experimental): Fixed dose ABBV-154 every other week.
  Interventions: Drug: ABBV-154
- Maintenance Phase: Randomized Placebo (Placebo Comparator): Fixed dose placebo every other week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABBV-154 — Intravenous (IV) Infusion; Subcutaneous Injection
  Arms: Induction Phase: ABBV-154 Randomized Dose A; Induction Phase: ABBV-154 Randomized Dose B; Induction Phase: ABBV-154 Randomized Dose C; Induction Phase: ABBV-154 Randomized Dose D; Re-Induction Phase: ABBV-154 Randomized Dose A; Re-Induction Phase: ABBV-154 Randomized Dose B
Drug: Placebo — Intravenous (IV) infusion; Subcutaneous Injection
  Arms: Induction Phase: Randomized Placebo
Drug: ABBV-154 — Subcutaneous Injection
  Arms: Maintenance Phase: ABBV-154 Randomized Dose A; Maintenance Phase: ABBV-154 Randomized Dose B
Drug: Placebo — Subcutaneous Injection
  Arms: Induction Phase: ABBV-154 Randomized Dose D; Maintenance Phase: Randomized Placebo

SUMMARY:
Crohn's disease (CD) is a long-lasting condition causing inflammation that can affect any part of the gut. CD may cause tiredness, loose stools with or without bleeding, abdominal pain, weight loss, and fever. This study evaluates how safe and effective ABBV-154 is in participants treated for moderately to severely active CD. Adverse events and change in the disease activity will be assessed.

ABBV-154 is an investigational drug being evaluated for the treatment of CD. In the induction period, there is a 1 in 5 chance that participants will be assigned to placebo. Depending on the dose received in the induction period, there is a 1 in 2 or 1 in 3 chance that participants will be assigned to placebo in the maintenance period. Around 265 participants 18-75 years of age with moderately to severely active CD will be enrolled in the study at approximately 200 sites worldwide.

The study is comprised of a 12-week double-blind, placebo-controlled induction period, followed by either a 12-week double-blind re-induction period for non-responders or a 40-week double-blind placebo-controlled maintenance period for responders. In the maintenance period, responders will be randomized to receive subcutaneous placebo or ABBV-154 in 2 different doses every other week. Participants in the placebo group who are initial responders will receive ABBV-154 in the maintenance period.

There may be higher treatment burden for participants in this trial compared to their standard of care due to study procedures. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Crohn's Disease (CD) for at least 3 months prior to Baseline of the Induction Period.
* Crohn's Disease Activity Index (CDAI) score 220 to 450 at Baseline of the Induction Period.
* Endoscopic evidence of mucosal inflammation as documented by an Simple Endoscopic Score for Crohn's Disease (SES-CD) of >= 6 for ileocolonic or colonic disease or SES-CD of >= 4 for isolated ileal disease as scored by a central reader. All eligible scores must exclude the presence of narrowing component.
* Demonstrated intolerance or inadequate response to one or more of the following biologic agents: infliximab, adalimumab, certolizumab pegol, vedolizumab, natalizumab, ustekinumab, or risankizumab.

Exclusion Criteria:

- Participants with prior intolerance to adalimumab.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (166):
- United States (45):
  - Digestive Health Specialists of the Southeast /ID# 239599, Dothan, Alabama
  - East View Medical Research, LLC /ID# 240030, Mobile, Alabama
  - Southern California Res. Ctr. /ID# 233512, Coronado, California
  - Hoag Memorial Hosp Presbyterian /ID# 233555, Irvine, California
  - University of Colorado Hospital /ID# 239361, Aurora, Colorado
  - Medical Research Center of CT /ID# 233542, Hamden, Connecticut
  - Atlantic Medical Research /ID# 233506, Margate, Florida
  - University of Miami /ID# 233811, Miami, Florida
  - Gastroenterology Group Naples /ID# 233829, Naples, Florida
  - Digestive Disease Consultants - Orange Park /ID# 241015, Orange Park, Florida
  - Endoscopic Research, Inc. /ID# 234279, Orlando, Florida
  - IMIC Inc. Medical Research /ID# 233821, Palmetto Bay, Florida
  - Emory University /ID# 241014, Atlanta, Georgia
  - AGILE Clinical Research Trials /ID# 233739, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, LLC /ID# 245604, Macon, Georgia
  - GI Specialists of GA, PC /ID# 239261, Marietta, Georgia
  - Gastroenterology Consultants, P.C /ID# 233552, Roswell, Georgia
  - The University of Chicago DCAM /ID# 233824, Chicago, Illinois
  - Digestive Health Services /ID# 241177, Downers Grove, Illinois
  - Southwest Gastroenterology /ID# 234278, Oak Lawn, Illinois
  - University of Louisville /ID# 233766, Louisville, Kentucky
  - Louisiana Research Center, LLC /ID# 245370, Shreveport, Louisiana
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 233765, Ann Arbor, Michigan
  - Gastroenterology Associates of Western Michigan, PLC d.b.a. West Michigan Clinic /ID# 233763, Wyoming, Michigan
  - Mayo Clinic - Rochester /ID# 238516, Rochester, Minnesota
  - Las Vegas Medical Research /ID# 233826, Las Vegas, Nevada
  - Allied Health Clinical Research Organization, LLC /ID# 241935, Englewood, New Jersey
  - The Mount Sinai Hospital /ID# 233823, New York, New York
  - Lenox Hill Hospital /ID# 239312, New York, New York
  - New York Gastroenterology Associates /ID# 241967, New York, New York
  - Univ NC Chapel Hill /ID# 233557, Chapel Hill, North Carolina
  - Northshore Gastroentrology Research LLC /ID# 239307, Brooklyn, Ohio
  - University of Cincinnati /ID# 234237, Cincinnati, Ohio
  - Hightower Clinical /ID# 239598, Oklahoma City, Oklahoma
  - Digestive Disease Specialists /ID# 233825, Oklahoma City, Oklahoma
  - University of Pennsylvania /ID# 239291, Philadelphia, Pennsylvania
  - Allegheny Health Network Research Institute /ID# 239334, Pittsburgh, Pennsylvania
  - Gastroenterology Associates, P.A. of Greenville /ID# 233544, Greenville, South Carolina
  - Gastro One /ID# 239748, Cordova, Tennessee
  - Southern Star Research Institute, LLC /ID# 240132, San Antonio, Texas
  - Tyler Research Institute, LLC /ID# 233730, Tyler, Texas
  - Gastro Health & Nutrition - Victoria /ID# 240158, Victoria, Texas
  - University of Utah Hospitals and Clinics /ID# 239264, Salt Lake City, Utah
  - Gastro Health Research /ID# 240085, Fairfax, Virginia
  - Hunter Holmes McGuire VA Medical Center /ID# 233759, Richmond, Virginia
- Australia (6):
  - Concord Repatriation General /ID# 233467, Concord, New South Wales
  - Princess Alexandra Hospital /ID# 234243, Woolloongabba, Queensland
  - Royal Adelaide Hospital /ID# 233705, Adelaide, South Australia
  - The Queen Elizabeth Hospital /ID# 234242, Woodville South, South Australia
  - Monash Medical Centre /ID# 233469, Clayton, Victoria
  - Fiona Stanley Hospital /ID# 240136, Murdoch, Western Australia
- Austria (3):
  - Medizinische Universitaet Innsbruck /ID# 234217, Innsbruck, Tyrol
  - Medizinische Universitaet Wien /ID# 234218, Vienna, Vienna
  - Landeskrankenhaus Salzburg-Universitätsklinikum der PMU (LKH) /ID# 234069, Salzburg
- Belgium (5):
  - UCL Saint-Luc /ID# 232435, Woluwe-Saint-Lambert, Brussels Capital
  - UZ Gent /ID# 246877, Ghent, Oost-Vlaanderen
  - AZ-Delta /ID# 232437, Roeselare, West-Vlaanderen
  - AZ Maria Middelares /ID# 246880, Ghent
  - CHU de Liege /ID# 232436, Liège
- Bulgaria (5):
  - UMHAT Kaspela /ID# 232468, Plovdiv
  - Second MHAT Sofia /ID# 250706, Sofia
  - UMHAT Sveti Ivan Rilski /ID# 233522, Sofia
  - UMHAT Tsaritsa Joanna - ISUL /ID# 234135, Sofia
  - Acibadem City Clinic University Hospital EOOD /ID# 240003, Sofia
- Canada (7):
  - University of Calgary /ID# 233838, Calgary, Alberta
  - Gastroenterology and Internal Medicine Research Institution /ID# 233831, Edmonton, Alberta
  - QE II Health Sciences Centre /ID# 233839, Halifax, Nova Scotia
  - London Health Sciences Center- University Hospital /ID# 234058, London, Ontario
  - Scott Shulman Medicine Professional Corporation /ID# 239567, North Bay, Ontario
  - Toronto Immune and Digestive Health Institute Inc /ID# 234142, North York, Ontario
  - Toronto Digestive Disease Associates, Inc. /ID# 234143, Vaughan, Ontario
- Czechia (4):
  - Hepato-Gastroenterologie HK, s.r.o. /ID# 239965, Hradec Králové
  - ARTROSCAN s.r.o. /ID# 239882, Ostrava
  - Nemocnice Horovice - NH Hospital a.s /ID# 233915, Prague
  - Ustredni Vojenska Nemocnice - Vojenska fakultni nemocnice Praha /ID# 238486, Prague
- France (4):
  - CHU Montpellier - Hôpital Saint Eloi /ID# 241136, Montpellier, Herault
  - CHRU Nancy - Hopitaux de Brabois /ID# 234224, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHU de SAINT ETIENNE - Hopital Nord /ID# 234225, Saint Priest EN Jarez, Pays de la Loire Region
  - AP-HP - Hopital Saint-Louis /ID# 234227, Paris
- Germany (10):
  - Universitaetsklinikum Freiburg /ID# 233719, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitatsklinikum Mannheim /ID# 233716, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 233531, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 233529, Erlangen, Bavaria
  - Universitatsklinik Regensburg /ID# 238702, Regensburg, Bavaria
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 233527, Kiel, Schleswig-Holstein
  - DRK Kliniken Berlin Westend /ID# 233718, Berlin
  - Medizinische Hochschule Hannover /ID# 238804, Hanover
  - EUGASTRO GmbH /ID# 233717, Leipzig
  - Klinikum Lueneburg /ID# 233720, Lüneburg
- Greece (4):
  - General Hospital of Athens Ippokratio /ID# 231655, Athens, Attica
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 231660, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 231657, Heraklion, Crete
  - General Hospital of Nikaia-Piraeus "Agios Panteleimon" /ID# 231659, Pireaus
- Clinfan Szolgaltato Kft. /ID# 249662, Szekszárd, Hungary
- Israel (6):
  - Shaare Zedek Medical Center /ID# 233460, Jerusalem, Jerusalem
  - Hadassah Medical Center-Hebrew University /ID# 233518, Jerusalem, Jerusalem
  - The Edith Wolfson Medical Center /ID# 234042, Ashkelon, Southern District
  - Soroka University Medical Center /ID# 233458, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 233457, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 238525, Tel Aviv, Tel Aviv
- Italy (4):
  - ASST Rhodense/Presidio Ospedaliero di Rho /ID# 233386, Rho, Milano
  - Policlinico Agostino Gemelli /ID# 233380, Rome, Roma
  - Azienda Ospedaliera Universitaria Consorziale Policlinico /ID# 233387, Bari
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 233382, Milan
- Japan (31):
  - Aichi Medical University Hospital /ID# 238528, Nagakute-shi, Aichi-ken
  - Daido Clinic /ID# 239730, Nagoya, Aichi-ken
  - Nagoya University Hospital /ID# 238662, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 238368, Nagoya, Aichi-ken
  - Tsujinaka Hospital Kashiwanoha /ID# 239012, Kashiwa-shi, Chiba
  - Fukushima Medical University Hospital /ID# 239314, Fukushima, Fukushima
  - Gunma University Hospital /ID# 239913, Maebashi, Gunma
  - Hiroshima University Hospital /ID# 238947, Hiroshima, Hiroshima
  - Asahikawa City Hospital /ID# 248061, Asahikawa-shi, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 238791, Sapporo, Hokkaido
  - Sapporo Medical University Hospital /ID# 239201, Sapporo, Hokkaido
  - Sapporo IBD Clinic /ID# 239054, Sapporo, Hokkaido
  - Hyogo Medical University Hospital /ID# 239049, Nishinomiya-shi, Hyōgo
  - Kanazawa University Hospital /ID# 239670, Kanazawa, Ishikawa-ken
  - Iwate Medical University Uchimaru Medical Center /ID# 238953, Morioka, Iwate
  - St. Marianna University Hospital /ID# 239167, Kawasaki-shi, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine /ID# 239918, Kyoto, Kyoto
  - Mie University Hospital /ID# 239758, Tsu, Mie-ken
  - Tohoku University Hospital /ID# 238476, Sendai, Miyagi
  - Okayama University Hospital /ID# 239757, Okayama, Okayama-ken
  - Osaka Metropolitan University Hospital /ID# 238638, Osaka, Osaka
  - Osaka University Hospital /ID# 240485, Suita-shi, Osaka
  - Hamamatsu University Hospital /ID# 238527, Hamamatsu, Shizuoka
  - NHO Shizuoka Medical Center /ID# 239759, Sunto-gun, Shizuoka
  - Tokyo Medical And Dental University Hospital /ID# 238950, Bunkyo-ku, Tokyo
  - Kyorin University Hospital /ID# 239609, Mitaka-shi, Tokyo
  - Tokyo Medical University Hospital /ID# 239668, Shinjuku-ku, Tokyo
  - Center hospital of the National Center for Global Health and Medicine /ID# 239792, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 239760, Shinjuku-ku, Tokyo
  - Japan Community Health care Organization Tokyo Yamate Medical Center /ID# 239554, Shinjuku-ku, Tokyo
  - Yamagata University Hospital /ID# 239572, Yamagata, Yamagata
- Netherlands (2):
  - Radboud Universitair Medisch Centrum /ID# 241292, Nijmegen, Gelderland
  - Academisch Medisch Centrum /ID# 232123, Amsterdam
- New Zealand (3):
  - Dunedin Hospital /ID# 238325, Otago, Otago
  - Wellington Regional Hospital /ID# 238326, Newtown, Wellington Region
  - Hutt Hospital /ID# 238327, Lower Hutt
- Poland (4):
  - Planetmed Sp. z o.o. /ID# 238447, Wroclaw, Lower Silesian Voivodeship
  - WIP Warsaw IBD Point Profesor Kierkus /ID# 233533, Warsaw, Masovian Voivodeship
  - Panstwowy Instytut Medyczny MSWiA w Warszawie /ID# 238653, Warsaw, Masovian Voivodeship
  - Endoskopia Sp. z o.o. /ID# 249906, Sopot, Pomeranian Voivodeship
- Portugal (2):
  - Hospital da Senhora da Oliveira Guimaraes, EPE /ID# 249047, Guimarães, Braga District
  - 2CA-Braga, Hospital de Braga /ID# 249049, Braga
- Mindful Medical Research /ID# 249609, San Juan, Puerto Rico
- Slovakia (3):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 232373, Banská Bystrica
  - ENDOMED s.r.o. /ID# 241855, Košice
  - KM Management, spol. s.r.o. /ID# 241849, Nitra
- South Korea (3):
  - The Catholic University of Korea, Daejeon St.Mary's Hospital /ID# 233700, Daejeon
  - Asan Medical Center /ID# 233701, Seoul
  - Samsung Medical Center /ID# 233698, Seoul
- Spain (4):
  - Hospital Arquitecto Marcide - Complejo Hospitalario Universitario de Ferrol /ID# 232299, Ferrol, A Coruna
  - Hospital Santa Creu i Sant Pau /ID# 232301, Barcelona
  - Hospital Universitario La Paz /ID# 232300, Madrid
  - Hospital Clinico Universitario de Valencia /ID# 234103, Valencia
- Taiwan (3):
  - China Medical University Hospital /ID# 234132, Taichung
  - Taichung Veterans General Hospital /ID# 234131, Taichung
  - National Taiwan University Hospital /ID# 234134, Taipei
- United Kingdom (6):
  - Royal Devon University Healthcare NHS Foundation Trust /ID# 234194, Exeter, Devon
  - University Hospital Southampton NHS Foundation Trust /ID# 238960, Southampton, Hampshire
  - Barts Health NHS Trust /ID# 234188, London, London, City of
  - Guys and St Thomas NHS Foundation Trust /ID# 234191, London, London, City of
  - NHS Greater Glasgow and Clyde /ID# 234186, Glasgow, Scotland
  - St George's University Hospitals NHS Foundation Trust /ID# 234193, Tooting

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this Double-Blind study, subjects with Crohn's Disease (CD) were randomized into 5 groups for 12 weeks (Induction Period). At week 12, subjects were categorized as responders or non-responders. Responders were re-randomized into a 40-Week Maintenance Period. Non-responders were re-randomized into the 12-Week Re-Induction Period. At week 12 of the re-induction period, those achieving clinical/endoscopic response were re-randomized into the Maintenance Period.
Groups:
- Placebo: Participants received Placebo Intravenous (IV) during Week (Wk) 0, followed by Placebo Subcutaneous (SC) Every Other Week (EOW) until week 12
  Maintenance Period:
  Participants received Placebo SC, EOW for 40 weeks
- ABBV-154 150mg IV, 80mg SC EOW: Participants received a loading dose of 150mg IV of ABBV-154 during Wk 0, followed by ABBV-154 80mg SC during Wk 2 and EOW until Week 12
- ABBV-154 300mg IV, 230mg SC EOW: Participants received 300mg IV of ABBV-154 during Wk 0, followed by ABBV-154 230mg SC during Wk 2 and EOW until Week 12
- ABBV-154 600mg IV, 530mg SC EOW: Participants received 600mg IV of ABBV-154 during Wk 0, followed by ABBV-154 530mg SC during Wk 2 and EOW until Week 12
- ABBV-154 600mg IV, 530mg SC E4W: Participants received 600mg IV of ABBV-154 during Wk 0, followed by ABBV-154 530mg SC during Wk 4 and Wk 8; every 4 weeks (E4W)
- ABBV-154 80mg SC EOW: During the Maintenance Period, participants received ABBV-154 80mg SC only. No IV was administered during the Maintenance Period.
- ABBV-154 230mg SC EOW: During the Maintenance Period, participants received ABBV-154 230mg SC only. No IV was administered during the Maintenance Period.
- MP: Placebo Responders; ABBV-154 80mg SC: During the Maintenance Period, placebo responders received ABBV-154 80mg SC only. No IV was administered during the Maintenance Period.
Period: Double-Blind Induction (12 Weeks)
Arm/Group | Placebo | ABBV-154 150mg IV, 80mg SC EOW | ABBV-154 300mg IV, 230mg SC EOW | ABBV-154 600mg IV, 530mg SC EOW | ABBV-154 600mg IV, 530mg SC E4W | ABBV-154 80mg SC EOW | ABBV-154 230mg SC EOW | MP: Placebo Responders; ABBV-154 80mg SC
Started | 21 | 20 | 22 | 20 | 23 | 0 | 0 | 0
Completed | 12 | 15 | 12 | 15 | 12 | 0 | 0 | 0
Not Completed | 9 | 5 | 10 | 5 | 11 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 7 | 2 | 6 | 5 | 10 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Period: Double-Blind Re-Induction (12 Weeks)
Arm/Group | Placebo | ABBV-154 150mg IV, 80mg SC EOW | ABBV-154 300mg IV, 230mg SC EOW | ABBV-154 600mg IV, 530mg SC EOW | ABBV-154 600mg IV, 530mg SC E4W | ABBV-154 80mg SC EOW | ABBV-154 230mg SC EOW | MP: Placebo Responders; ABBV-154 80mg SC
Started | 0 | 0 | 12 | 12 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 9 | 6 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 3 | 6 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Period: Double-Blind Maintenance (40 Weeks)
Arm/Group | Placebo | ABBV-154 150mg IV, 80mg SC EOW | ABBV-154 300mg IV, 230mg SC EOW | ABBV-154 600mg IV, 530mg SC EOW | ABBV-154 600mg IV, 530mg SC E4W | ABBV-154 80mg SC EOW | ABBV-154 230mg SC EOW | MP: Placebo Responders; ABBV-154 80mg SC
Started | 18 | 0 | 0 | 0 | 0 | 14 | 13 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 18 | 0 | 0 | 0 | 0 | 13 | 13 | 4
Not completed — Lack of efficacy w/o receiving ABBV-154 rescue | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor after ABBV-154 | 8 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Not completed — AE w/o receiving ABBV-154 rescue | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — WD by subject w/o receiving ABBV-154 rescue | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of efficacy after receiving ABBV-154 rescue | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor w/o receiving ABBV-154 rescue | 6 | 0 | 0 | 0 | 0 | 10 | 11 | 3
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT1 population; all enrolled
Groups:
- Double-Blind Induction Phase: Placebo: Fixed dose placebo as described in the protocol.
  Placebo: Intravenous (IV) infusion; Subcutaneous Injection.
- Double-Blind Induction Phase: ABBV-154 150mg IV/ 80mg SC EOW: ABBV-154:
  150 mg Intravenous (IV) Infusion and Subcutaneous Injection 80 mg (SC) at end of week (EOW) 12-week double-blind Induction Phase.
- Double-Blind Induction Phase: ABBV-154 300mg IV/ 230mg SC EOW: ABBV-154:
  300 mg Intravenous (IV) Infusion and Subcutaneous Injection 230 mg (SC) at end of week (EOW) 12-week double-blind Induction Phase.
- Double-Blind Induction Phase: ABBV-154 600mg IV/ 530mg SC EOW: ABBV-154:
  600 mg Intravenous (IV) Infusion and Subcutaneous Injection 530 mg (SC) at end of week (EOW) 12-week double-blind Induction Phase.
- Double-Blind Induction Phase: ABBV-154 600mg IV/ 530mg SC E4W: ABBV-154:
  600 mg Intravenous (IV) Infusion and Subcutaneous Injection 530 mg (SC) every 4 weeks (E4W) 12-week double-blind Induction Phase.
- Total: Total of all reporting groups
Arm/Group | Double-Blind Induction Phase: Placebo | Double-Blind Induction Phase: ABBV-154 150mg IV/ 80mg SC EOW | Double-Blind Induction Phase: ABBV-154 300mg IV/ 230mg SC EOW | Double-Blind Induction Phase: ABBV-154 600mg IV/ 530mg SC EOW | Double-Blind Induction Phase: ABBV-154 600mg IV/ 530mg SC E4W | Total
Number analyzed (Participants) | 21 | 20 | 22 | 20 | 23 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (13.23) | 41.7 (14.27) | 39.6 (12.23) | 43.1 (14.37) | 42.0 (14.20) | 41.0 (13.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 8 | 9 | 10 | 43
  Male | 13 | 12 | 14 | 11 | 13 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 21 | 20 | 21 | 20 | 23 | 105
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 5 | 4 | 5 | 4 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 2 | 3
  White | 17 | 15 | 17 | 14 | 17 | 80
  More than one race | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Baseline Simple Endoscopic Score for Crohn's Disease (SES-CD) for ITT1 (all enrolled) [Mean (Standard Deviation); unit: SES-CD score (0-56)] — ITT1 population; all enrolled. Note: Percentages calculated on non-missing values. The SES-CD evaluates 4 endoscopic variables (ulcer size, ulcerated surface, affected surface, and narrowing, each on a scale from 0 (none) to 3 (worst) in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, sigmoid and left colon, and rectum). The total score is the sum of the 4 endoscopic variable scores and ranges from 0 to 56, where higher scores indicate more severe disease.
  SES-CD score (0-56) | 14.86 (8.928) | 13.53 (6.816) | 16.73 (10.533) | 16.13 (6.472) | 14.65 (6.748) | 15.19 (8.011)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Endoscopic Response Per Simple Endoscopic Score for Crohn's Disease (SES-CD)
Description: The SES-CD assesses endoscopic disease severity by evidence of active intestinal mucosal inflammation. Endoscopic response is defined as a decrease in SES-CD > 50% from Baseline (or for participants with isolated ileal disease and a Baseline SES-CD of 4, at least a 2-point reduction from Baseline). The SES-CD evaluates 4 endoscopic variables (ulcer size, ulcerated surface, affected surface, and narrowing, each on a scale from 0 (none) to 3 (worst) in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, sigmoid and left colon, and rectum). The total score is the sum of the 4 endoscopic variable scores and ranges from 0 to 56, where higher scores indicate more severe disease.
Time Frame: Baseline to Week 12
Population: ITT1 Population for whom data was collected and available for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants received Placebo Intravenous (IV) during Week (Wk) 0, followed by Placebo Subcutaneous (SC) Every Other Week (EOW) until week 12
- ABBV-154 150mg IV, 80mg SC EOW: Participants received 150mg IV of ABBV-154 during Wk 0, followed by ABBV-154 80mg SC during Wk 2 and EOW until Week 12
Arm/Group | Placebo | ABBV-154 150mg IV, 80mg SC EOW | ABBV-154 300mg IV, 230mg SC EOW | ABBV-154 600mg IV, 530mg SC EOW | ABBV-154 600mg IV, 530mg SC E4W
Number analyzed (Participants) | 11 | 14 | 12 | 14 | 11
Participants | 0 | 1 | 4 | 4 | 3
Statistical Analysis 1: Comparison: Placebo vs ABBV-154 150mg IV, 80mg SC EOW; Test type: Superiority; Risk Difference (RD) = 7.1, 95% CI 2-sided [-6.3 to 20.6] — Risk difference = (ABBV-154 - placebo)
Statistical Analysis 2: Comparison: Placebo vs ABBV-154 300mg IV, 230mg SC EOW; Test type: Superiority; Risk Difference (RD) = 33.3, 95% CI 2-sided [6.7 to 60.0] — Risk difference = (ABBV-154 - placebo)
Statistical Analysis 3: Comparison: Placebo vs ABBV-154 600mg IV, 530mg SC EOW; Test type: Superiority; Risk Difference (RD) = 28.6, 95% CI 2-sided [4.9 to 52.2] — Risk difference = (ABBV-154 - placebo)
Statistical Analysis 4: Comparison: Placebo vs ABBV-154 600mg IV, 530mg SC E4W; Test type: Superiority; Risk Difference (RD) = 27.3, 95% CI 2-sided [1.0 to 53.6] — Risk difference = (ABBV-154 - placebo)

2. Secondary Outcome: Percentage of Participants Achieving Clinical Remission Per Crohn's Disease Activity Index (CDAI)
Description: The CDAI consists of 8 components; 6 are based on participant diary entries, participant interviews, and physical examinations, and 2 are based on laboratory analysis, and measurement of body weight and height. Clinical remission is defined as CDAI < 150.
Time Frame: Induction Period Week 12
Population: ITT1 Population for whom data was collected and available for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- ABBV-154 150mg IV/ 80mg SC EOW: Participants received 150mg IV of ABBV-154 during Wk 0, followed by ABBV-154 80mg SC during Wk 2 and EOW until Week 12
- ABBV-154 300mg IV/ 230mg SC EOW: Participants received 300mg IV of ABBV-154 during Wk 0, followed by ABBV-154 230mg SC during Wk 2 and EOW until Week 12
- ABBV-154 600mg IV/ 530mg SC EOW: Participants received 600mg IV of ABBV-154 during Wk 0, followed by ABBV-154 530mg SC during Wk 2 and EOW until Week 12
- ABBV-154 600mg IV/ 530mg SC E4W: Participants received 600mg IV of ABBV-154 during Wk 0, followed by ABBV-154 530mg SC during Wk 4 and Wk 8; every 4 weeks (E4W)
Arm/Group | Placebo | ABBV-154 150mg IV/ 80mg SC EOW | ABBV-154 300mg IV/ 230mg SC EOW | ABBV-154 600mg IV/ 530mg SC EOW | ABBV-154 600mg IV/ 530mg SC E4W
Number analyzed (Participants) | 12 | 14 | 13 | 14 | 10
Participants | 2 | 4 | 6 | 5 | 4
Statistical Analysis 1: Comparison: Placebo vs ABBV-154 150mg IV/ 80mg SC EOW; Test type: Superiority; Risk Difference (RD) = 11.9, 95% CI 2-sided [-19.8 to 43.6] — Risk difference = (ABBV-154 - placebo)
Statistical Analysis 2: Comparison: Placebo vs ABBV-154 300mg IV/ 230mg SC EOW; Test type: Superiority; Risk Difference (RD) = 29.5, 95% CI 2-sided [-4.8 to 63.8] — Risk difference = (ABBV-154 - placebo)
Statistical Analysis 3: Comparison: Placebo vs ABBV-154 600mg IV/ 530mg SC EOW; Test type: Superiority; Risk Difference (RD) = 19.0, 95% CI 2-sided [-13.7 to 51.8] — Risk difference = (ABBV-154 - placebo)
Statistical Analysis 4: Comparison: Placebo vs ABBV-154 600mg IV/ 530mg SC E4W; Test type: Superiority; Risk Difference (RD) = 23.3, 95% CI 2-sided [-13.6 to 60.3] — Risk difference = (ABBV-154 - placebo)

3. Secondary Outcome: Percentage of Participants Achieving Clinical Remission Per Average Daily Liquid or Very Soft Stool Frequency (SF) and Average Daily Abdominal Pain (AP) Score (SF/AP)
Description: Clinical remission is defined as average daily liquid or very soft stool SF <= 2.8 and not worse than Baseline and average daily AP score <= 1 and not worse than Baseline.
Time Frame: Induction Period Week 12
Population: ITT1 Population for whom data was collected and available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ABBV-154 150mg IV, 80mg SC EOW | ABBV-154 300mg IV, 230mg SC EOW | ABBV-154 600mg IV, 530mg SC EOW | ABBV-154 600mg IV, 530mg SC E4W
Number analyzed (Participants) | 13 | 15 | 13 | 15 | 11
Participants | 2 | 4 | 7 | 6 | 6
Statistical Analysis 1: Comparison: Placebo vs ABBV-154 150mg IV, 80mg SC EOW; Test type: Superiority; Risk Difference (RD) = 11.3, 95% CI 2-sided [-18.5 to 41.0] — Risk difference = (ABBV-154 - placebo)
Statistical Analysis 2: Comparison: Placebo vs ABBV-154 300mg IV, 230mg SC EOW; Test type: Superiority; Risk Difference (RD) = 38.5, 95% CI 2-sided [5.0 to 71.9] — Risk difference = (ABBV-154 - placebo)
Statistical Analysis 3: Comparison: Placebo vs ABBV-154 600mg IV, 530mg SC EOW; Test type: Superiority; Risk Difference (RD) = 24.6, 95% CI 2-sided [-7.0 to 56.2] — Risk difference = (ABBV-154 - placebo)
Statistical Analysis 4: Comparison: Placebo vs ABBV-154 600mg IV, 530mg SC E4W; Test type: Superiority; Risk Difference (RD) = 39.2, 95% CI 2-sided [3.8 to 74.5] — Risk difference = (ABBV-154 - placebo)

4. Secondary Outcome: Percentage of Participants Achieving Endoscopic Response Per SES-CD
Description: The SES-CD assesses endoscopic disease severity by evidence of active intestinal mucosal inflammation. Endoscopic response is defined as a decrease in SES-CD > 50% from Baseline (or for participants with isolated ileal disease and a Baseline SES-CD of 4, at least a 2-point reduction from Baseline).
Time Frame: Week 40 in the Maintenance Period
Population: Data were not collected for this outcome due to early termination of the study.
Arm/Group | Placebo | ABBV-154 80mg SC EOW | ABBV-154 230mg SC EOW
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants Achieving Clinical Remission Per CDAI
Description: as for outcome 2
Time Frame: Week 40 in the Maintenance Period
Population: Data were not collected for this outcome due to early termination of the study.
Arm/Group | Placebo | ABBV-154 80mg SC EOW | ABBV-154 230mg SC EOW
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants Achieving Clinical Remission Per SF/AP
Description: Clinical remission is defined as average daily liquid or very soft SF <= 2.8 and not worse than Baseline and average daily AP score <= 1 and not worse than Baseline.
Time Frame: Week 40 in the Maintenance Period
Population: Data were not collected for this outcome due to early termination of the study.
Arm/Group | Placebo | ABBV-154 80mg SC EOW | ABBV-154 230mg SC EOW
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality were reported from enrollment to study termination, median time on follow up was 85 days(d) for Placebo and ABBV-154 150 IV/80 SC; 87.5d for ABBV-154 300 IV/230 SC; 86d for ABBV-154 600 IV/ 530 SC; and 84d for ABBV-154 600 IV/ 530 SC E4W. Treatment-emergent and serious AE were collected from first dose until 70d after last dose; mean duration on study drug was 12 weeks for each group.
Groups:
- Induction Period: Placebo: Participants received Placebo Intravenous (IV) during Week (Wk) 0, followed by Placebo Subcutaneous (SC) Every Other Week (EOW) until week 12
- Induction Period: ABBV-154 150mg IV, 80mg SC: Participants received 150mg IV of ABBV-154 during Wk 0, followed by ABBV-154 80mg SC during Wk 2 and EOW until Week 12
- Induction Period: ABBV-154 300mg IV, 230mg SC: Participants received 300mg IV of ABBV-154 during Wk 0, followed by ABBV-154 230mg SC during Wk 2 and EOW until Week 12
- Induction Period: ABBV-154 600mg IV, 530mg SC: Participants received 600mg IV of ABBV-154 during Wk 0, followed by ABBV-154 530mg SC during Wk 2 and EOW until Week 12
- Induction Period: ABBV-154 600mg IV, 530mg SC E4W: Participants received 600mg IV of ABBV-154 during Wk 0, followed by ABBV-154 530mg SC during Wk 4 and Wk 8; every 4 weeks (E4W)
- IP: Placebo; ReIP: ABBV-154 300mg IV, 230mg SC: Following Induction Period (IP): Non-responding, Placebo-dosed Participants were re-induced (ReIP) with ABBV-154 300mg IV (Wk 12), followed by 230mg SC (Wk 14) and EOW until Wk 24
- IP: Placebo; ReIP: ABBV-154 600mg IV, 530mg SC: Following IP: Non-responding, Placebo-dosed Participants were ReIP with ABBV-154 600mg IV (Wk 12), followed by 530mg SC (Wk 14) and EOW until Wk 24
- IP: ABBV-154; ReIP: ABBV-154 300mg IV, 230mg SC: Following IP: Non-responding, ABBV-154-dosed Participants were ReIP with ABBV-154 300mg IV (Wk 12), followed by 230mg SC (Wk 14) and EOW until Wk 24
- IP: ABBV-154; ReIP: ABBV-154 600mg IV, 530mg SC: Following IP: Non-responding, ABBV-154-dosed Participants were ReIP with ABBV-154 600mg IV (Wk 12), followed by 530mg SC (Wk 14) and EOW until Wk 24
- MP: ABBV-154 Responders; Placebo SC: Following IP: Responding, ABBV-154-dosed Participants received Placebo SC EOW during the maintenance period (MP) of 40 weeks
- MP: ABBV-154 Responders; ABBV-154 80mg SC: Following IP: Responding, ABBV-154-dosed Participants received ABBV-154 80mg SC EOW during the maintenance period (MP) of 40 weeks
- MP: ABBV-154 Responders; ABBV-154 230mg SC: Following IP: Responding, ABBV-154-dosed Participants received ABBV-154 230mg SC EOW during the maintenance period (MP) of 40 weeks
- MP: Placebo Responders; ABBV-154 80mg SC: Following IP: Responding, Placebo-dosed Participants received ABBV-154 80mg SC EOW during the maintenance period (MP) of 40 weeks
- Rescue ABBV-154 600mg IV, 230mg SC EOW: During MP:
  Inadequate-Responding, Placebo or ABBV-154-dosed Participants received ABBV-154 600mg IV followed by 230mg SC Rescue Therapy
Arm/Group | Induction Period: Placebo | Induction Period: ABBV-154 150mg IV, 80mg SC | Induction Period: ABBV-154 300mg IV, 230mg SC | Induction Period: ABBV-154 600mg IV, 530mg SC | Induction Period: ABBV-154 600mg IV, 530mg SC E4W | IP: Placebo; ReIP: ABBV-154 300mg IV, 230mg SC | IP: Placebo; ReIP: ABBV-154 600mg IV, 530mg SC | IP: ABBV-154; ReIP: ABBV-154 300mg IV, 230mg SC | IP: ABBV-154; ReIP: ABBV-154 600mg IV, 530mg SC | MP: ABBV-154 Responders; Placebo SC | MP: ABBV-154 Responders; ABBV-154 80mg SC | MP: ABBV-154 Responders; ABBV-154 230mg SC | MP: Placebo Responders; ABBV-154 80mg SC | Rescue ABBV-154 600mg IV, 230mg SC EOW
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/22 | 0/20 | 0/23 | 0/4 | 0/4 | 0/8 | 0/8 | 0/18 | 0/14 | 0/13 | 0/4 | 0/14
Serious Adverse Events (participants affected / at risk) | 3/21 | 3/20 | 2/22 | 0/20 | 3/23 | 0/4 | 0/4 | 1/8 | 2/8 | 3/18 | 1/14 | 0/13 | 0/4 | 1/14
Other Adverse Events (participants affected / at risk) | 7/21 | 12/20 | 11/22 | 14/20 | 13/23 | 4/4 | 1/4 | 5/8 | 4/8 | 9/18 | 10/14 | 8/13 | 2/4 | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Period: Placebo (N=21) | Induction Period: ABBV-154 150mg IV, 80mg SC (N=20) | Induction Period: ABBV-154 300mg IV, 230mg SC (N=22) | Induction Period: ABBV-154 600mg IV, 530mg SC (N=20) | Induction Period: ABBV-154 600mg IV, 530mg SC E4W (N=23) | IP: Placebo; ReIP: ABBV-154 300mg IV, 230mg SC (N=4) | IP: Placebo; ReIP: ABBV-154 600mg IV, 530mg SC (N=4) | IP: ABBV-154; ReIP: ABBV-154 300mg IV, 230mg SC (N=8) | IP: ABBV-154; ReIP: ABBV-154 600mg IV, 530mg SC (N=8) | MP: ABBV-154 Responders; Placebo SC (N=18) | MP: ABBV-154 Responders; ABBV-154 80mg SC (N=14) | MP: ABBV-154 Responders; ABBV-154 230mg SC (N=13) | MP: Placebo Responders; ABBV-154 80mg SC (N=4) | Rescue ABBV-154 600mg IV, 230mg SC EOW (N=14)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLAMMATION (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED HYPERSENSITIVITY REACTION (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SERUM SICKNESS (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLONIC ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FOCAL PERITONITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Period: Placebo (N=21) | Induction Period: ABBV-154 150mg IV, 80mg SC (N=20) | Induction Period: ABBV-154 300mg IV, 230mg SC (N=22) | Induction Period: ABBV-154 600mg IV, 530mg SC (N=20) | Induction Period: ABBV-154 600mg IV, 530mg SC E4W (N=23) | IP: Placebo; ReIP: ABBV-154 300mg IV, 230mg SC (N=4) | IP: Placebo; ReIP: ABBV-154 600mg IV, 530mg SC (N=4) | IP: ABBV-154; ReIP: ABBV-154 300mg IV, 230mg SC (N=8) | IP: ABBV-154; ReIP: ABBV-154 600mg IV, 530mg SC (N=8) | MP: ABBV-154 Responders; Placebo SC (N=18) | MP: ABBV-154 Responders; ABBV-154 80mg SC (N=14) | MP: ABBV-154 Responders; ABBV-154 230mg SC (N=13) | MP: Placebo Responders; ABBV-154 80mg SC (N=4) | Rescue ABBV-154 600mg IV, 230mg SC EOW (N=14)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CUSHING'S SYNDROME (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
APHTHOUS ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 2 (2) | 2 (2)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHOIDS THROMBOSED (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PROCTALGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
FEELING ABNORMAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE BRUISING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE DRYNESS (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE ERYTHEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
INJECTION SITE EXFOLIATION (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE INDENTATION (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE PRURITUS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INJECTION SITE RASH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INJECTION SITE SWELLING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
LIVER DISORDER (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED HYPERSENSITIVITY REACTION (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
CRYPTOSPORIDIOSIS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ESCHERICHIA INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GINGIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PARONYCHIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RECTAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SALMONELLOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TINEA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIRAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CLOSTRIDIUM TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FAECAL CALPROTECTIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INCREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TENDON PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OPHTHALMIC MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PROSTATOMEGALY (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS PSORIASIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYTHROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LICHENOID KERATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH VESICULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
AbbVie has decided to discontinue further subject enrollment in the M20-371 (ABBV-154) study. This decision is not based on a safety or an efficacy signal; rather this decision was made because of a change in AbbVie's development.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT05068284/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT05068284/SAP_001.pdf